CLINICAL TRIAL: NCT01209533
Title: Inhaled Iloprost in Mild Asthma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Actelion (Industry)
Responsible Party: J.R. Sheller, M.D., Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 100637
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Iloprost — Inhaled iloprost 2.5 or 5 micrograms four times daily for 14 days
  Other Names: Ventavis

SUMMARY:
The purpose of the study is to determine if inhaled iloprost given four times daily can improve symptoms and lung function in adults with mild asthma.

DETAILED DESCRIPTION:
Animal studies have suggested that prostacyclin may downregulate allergic inflammation, thus providing the scientific basis for trials of inhaled prostacyclin agonists such as iloprost for the treatment of asthma. This study will examine the tolerability of four times daily iloprost on asthma symptoms and pulmonary function over a two week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60
2. History of asthma controlled by inhaled rescue medication (albuterol, levalbuterol etc) and/or inhaled corticosteroids
3. Ability to give informed consent
4. Ability to perform pulmonary function tests
5. Ability to tolerate the initial Ventavis inhalation
6. Ability to comply with the study protocol

Exclusion Criteria:

1. Cigarette smoking
2. Concomitant serious disease such as diabetes, hypertension, coronary heart disease, other lung disease, cancer (other than skin cancer)
3. Pregnancy or lack of contraception (hormonal or barrier)
4. Allergies or intolerance to inhaled iloprost
5. Participation in other ongoing research studies
6. Any psychological problem that the investigators believe might interfere with the conduct of the investigation.
7. Cigarette smoking
8. History of bleeding disorder, use of anticoagulants
9. Viral upper respiratory tract infection within the last 6 weeks
10. Table of upper limit for steroid use Beclomethasone dipropionate HFA-MDI 480 Budesonide DPI 1200 Flunisolide HFA-MDI 640 Fluticasone HFA-MDI 440 Fluticasone DPI 500 Mometasone DPI 440 Triamcinolone 1500 (Table adapted from EPR3, daily doses are in micrograms) Asthmatics requiring higher doses of inhaled corticosteroids than those given above, or using oral steroids, leukotriene modifiers, mast cell stabilizers, omalizumab, theophylline or long acting beta agonists will be excluded.
11. .Any screening laboratory blood test value outside the normal range will exclude the individual from the study, though an isolated abnormal value could be retested at an interval of no less than a week.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
PD20FEV1 methacholine | two weeks
  Provocative dose of methacholine resulting in a 20% fall in FEV1 from baseline

SECONDARY OUTCOMES:
asthma related symptoms | 4 weeks
  Asthma quality of life questionnaire; Juniper
asthma control | 4wks
  Juniper asthma control test score
FEV1 | 2wks
  Forced expiratory flow in one second
Exhaled nitric oxide | 2 wks
  Measurement of exhaled nitric oxide
Interleukin 17 | 2wks
  ELISA measurement of serum interleukin 17

CONTACTS AND LOCATIONS:
Overall Officials: James Sheller, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States